CLINICAL TRIAL: NCT02441517
Title: A Multicenter, Open-label, Single-arm, Study of Enzalutamide Re-Treatment in Metastatic Castration-Resistant Prostate Cancer, As First Treatment Post-Chemotherapy in Patients Who Have Previously Received Enzalutamide in the Pre-Chemotherapy Setting
Brief Title: A Study of Enzalutamide Re-treatment in Metastatic Castration-resistant Prostate Cancer After Docetaxel and/or Cabazitaxel Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study is closed early due to lck of enrollment.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-MA-1008
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Xtandi; Metastatic Castration Resistant Prostate Cancer; Metastatic; Prostate Cancer; Chemotherapy; Castration-resistant; Enzalutamide
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enzalutamide (Experimental): Participants received 160 mg enzalutamide orally once daily until radiographic or clinical progression, or unacceptable toxicity.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Participants were administered four 40-mg capsules orally once daily and taken as close to the same time each day as possible and could be taken with or without food.
  Other Names: ASP9785; Xtandi; MDV3100

SUMMARY:
The purpose of the study was to understand if there is benefit in treatment with a medicine called enzalutamide in the re-treatment setting. Patients must have been previously treated with enzalutamide in the pre-chemotherapy setting for a minimum of 8 months and have disease progressed, followed by docetaxel and/or cabazitaxel for at least 4 cycles.

DETAILED DESCRIPTION:
Participants received treatment with open-label enzalutamide, until radiographic or clinical progression (such as pathological fracture, cord compression, worsened pain requiring radiation therapy, or opioid analgesic dose increase or initiation), or unacceptable toxicity. Participants were to be allowed to continue enzalutamide until the next treatment was initiated. If another non-cytotoxic, non-investigational, antineoplastic agent was initiated after protocol-defined progression had been determined, enzalutamide was to be continued as long as the participant was tolerating enzalutamide and continued androgen deprivation therapy. Participants were to have a safety follow-up visit approximately 30 days following the last dose of study drug or prior to the initiation of a subsequent anti-cancer drug or investigational agent, whichever occurred first. Disease progression and survival were to be followed every 12 weeks for a maximum of 3 years from first dose. The study should have ended when the last participant has been followed for 1 year from the date of first dose, but the study was terminated and results up to the last date of evaluation (15 March 2017) are reflected in this disclosure.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without signet ring cell features.
* Presence of metastatic disease (M1) as assessed by computed tomography/ magnetic resonance imaging (CT/MRI) and/or whole-body radionuclide bone scan.
* Subject has been previously treated with enzalutamide for at least 8 months, and stopped enzalutamide due to progressive disease (not due to adverse events), followed by at least 4 cycles of docetaxel and/or cabazitaxel chemotherapy, with or without other intervening anti-cancer therapies (including but not limited to aminoglutethimide, ketoconozole, abiraterone acetate, Rad-223, or sipuleucel-T), prior to receiving chemotherapy. Note: for patients who receive sequential taxanes, there must not have been progressive disease upon ending the first taxane, or use of any anti-cancer agents between the two taxanes.
* Ongoing androgen deprivation therapy with an gonadotropin releasing hormone (GnRH) analogue or prior bilateral orchiectomy (medical or surgical castration). For patients who have not had bilateral orchiectomy, there must be a plan to maintain effective GnRH-analogue for the duration of the trial.
* Testosterone ≤ 1.73 nmol/L (≤ 50 ng/dL) at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at screening.
* Estimated life expectancy of ≥ 6 months at screening.
* Ability to swallow study drugs and to comply with study requirements throughout the study.
* Throughout study, male subject and a female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration. Two acceptable methods of birth control thus include the following:

  * Condom (barrier method of contraception) AND
  * One of the following is required:
  * Established use of oral, injected, or implanted hormonal method of contraception by the female partner performed at least 6 months before screening;
  * Placement of an intrauterine device or intrauterine system by the female partner;
  * Additional barrier method: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female partner;
  * Tubal ligation in the female partner.
  * Vasectomy or other procedure resulting in infertility (e.g., bilateral orchiectomy), performed at least 6 months before screening
* Must not donate sperm from screening through 3 months after final study drug administration.

Exclusion Criteria:

* Known or suspected neuroendocrine/small cell feature.
* Use of any antineoplastic treatment post-chemotherapy, including but not limited to aminoglutethimide, ketoconozole, abiraterone acetate, Rad-223, sipuleucel-T, or enzalutamide. Continuing steroids is permitted.
* Palliative radiation therapy within 2 weeks of Day 1, or within 4 weeks of Day 1 if a radionuclide was utilized.
* Use of an investigational agent within 4 weeks of Day 1 visit.
* Major surgery within 4 weeks prior to Day 1 visit.
* History of seizure or any condition that may predispose to seizures (e.g., prior cortical stroke or significant brain trauma) at any time in the past. History of loss of consciousness or transient ischemic attack within 12 months of screening.
* History of clinically significant cardiovascular disease including:

  * Myocardial infarction or uncontrolled angina within 3 months;
  * History of congestive heart failure New York Heart Association (NYHA) class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within three months results in a left ventricular ejection fraction that is ≥ 45%;
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place.
* Clinically significant cardiovascular disease at screening including:

  * Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mm Hg) at screening;
  * Bradycardia as indicated by a heart rate of < 45 beats per minute on the screening electrocardiogram (ECG) and on physical examination;
  * Uncontrolled hypertension as indicated by at least 2 consecutive measurements of a resting systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the screening visit.
* Subject has a known or suspected hypersensitivity to enzalutamide or any components of the formulation used.
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment.
* Known or suspected brain metastasis or leptomeningeal disease.
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months).
* Absolute neutrophil count < 1,500/μL, platelet count < 75,000/μL, or hemoglobin < 5.6 mmol/L (9 g/dL) at screening.
* Total bilirubin or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 times upper limit of normal (ULN) at screening.
* Creatinine > 177 μmol/L (> 2 mg/dL) at screening.
* Albumin < 30 g/L (3.0 g/dL) at screening.
* Treatment with abiraterone acetate prior to enzalutamide for metastatic castration - resistant prostate cancer (mCRPC) in the prechemotherapy setting. (Note: Patients who have received concomitant enzalutamide and abiraterone acetate therapies are not excluded).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Oncology, Study Director — APGD, Medical Affairs, Americas
Locations (5):
- United States (5):
  - Site US10003, Evanston, Illinois
  - Site US10006, Worcester, Massachusetts
  - Site US10004, New York, New York
  - Site US10001, Charleston, South Carolina
  - Site US10002, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male participants from the United States were enrolled in this study.
Pre-assignment Details: Metastatic castration-resistant prostate cancer (mCRPC) patients who were previously treated with enzalutamide (for a minimum of 8 months), followed by docetaxel and/or cabazitaxel chemotherapy (for a minimum of 4 cycles) were enrolled in this study.
Period: Overall Study
Arm/Group | Enzalutamide
Started | 4
Received Treatment | 4
Completed | 0
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was the safety analysis set (SAF), which consisted of all participants who took at least one dose of study medication.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Any Prior Radiotherapy [Count of Participants; unit: Participants]
  Yes | 2
  No | 2
Any Prior Disease-Related Surgeries [Count of Participants; unit: Participants]
  Yes | 2
  No | 2

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (rPFS)
Description: Radiographic PFS (rPFS) was defined as the time from first dose to the radiographic disease progression (PD), or death on study, whichever occurred first. Radiological PD was defined by either soft tissue tumor progression defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, or bone progression defined by the Prostate Cancer Clinical Trials Working Group 2 (PCWG2). Bone progression per PCWG2 was defined as a minimum of two new lesions. Progression on bone scans at time points before or at week 9 required a confirmatory scan performed six or more weeks later, where it should have demonstrated at least 2 additional new lesions (PCWG2) compared to the week 9 scan. rPFS was analyzed using Kaplan-Meier methodology to account for censored outcomes (i.e., no observation of rPFS event within the study follow-up period).
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the full analysis set (FAS), which consisted of all participants who are enrolled in the study, received at least one dose of study drug, and have at least one post baseline evaluation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 4
days | 115 [57 to 173]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the date of death due to any cause minus the date of first dose + 1.
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the FAS. Only participants with an overall survival event were included in the analysis.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: The time to PSA progression was defined as the PSA progression date minus the date of first dose + 1. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir (lowest PSA value observed postbaseline or the baseline value for participants who did not have a decline in PSA postbaseline values) in PSA levels, and which was confirmed by a second consecutive value obtained at least 3 or more weeks later (i.e., a confirmed rising trend) (PCWG2 criteria). The date of PSA progression was the first date the PSA progression was observed. Time to PSA progression was estimated via Kaplan-Meier methodology with censoring defined by the time of the last available PSA measure.
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 4
days | 82.5 [1 to 142]

4. Secondary Outcome: Number of Participants With PSA Response
Description: PSA response was defined for the three following categories: PSA30 response: a maximum decline of ≥ 30% from baseline at any post baseline time point; PSA50 response: a maximum decline of ≥ 50% from baseline at any post baseline time point; PSA90 response: a maximum decline of ≥ 90% from baseline at any post baseline time point.
Time Frame: From baseline up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the FAS. Only participants with at least 1 postbaseline PSA measure were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 4
Participants
  PSA30 Response | 2
  PSA50 Response | 2
  PSA90 Response | 0

5. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response was defined as the best overall response of complete response (CR) or partial response (PR) per RECIST 1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the FAS. Only participants with measurable disease at baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 4
Participants
  Complete Response | 0
  Partial Response | 0

6. Secondary Outcome: Time to First Use of a Subsequent Antineoplastic Therapy
Description: Time to start of other antineoplastic therapy was defined as the date of the first systemic antineoplastic therapy minus the date of the first dose of study drug + 1.
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the FAS. Only participants who underwent subsequent antineoplastic therapy were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 1
days | 175 [NA to NA] — Data could not be calculated as there were only 1 participant who had antineoplastic therapy.

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety was assessed by adverse events (AEs), which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE (SAE) was an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. Disease progression was not to be reported as an AE, and clinical signs and symptoms due to disease progression were collected as AEs.
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Population: The analysis population was the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 4
Participants
  Any TEAE | 4
  Drug-related TEAEs | 3
  Deaths | 0
  SAEs | 0
  Drug-related SAEs | 0
  Deaths Resulting from TEAEs | 0
  TEAEs Leading to Permanent Discontinuation | 0
  Drug-related TEAEs Leading to Permanent Discont. | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to date of last evaluation of 15 March 2017 (approximately 17 months)
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=4)
Fatigue (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hot flush (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT02441517/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02441517/SAP_001.pdf